CLINICAL TRIAL: NCT04809142
Title: A Randomized, Open-label, Parallel Controlled, Multi-center Phase III Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule Versus Chemotherapy as Second-line Treatment in Subjects With Advanced Biliary Cancer
Brief Title: A Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule as Second-line Treatment in Subjects With Advanced Biliary Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-III-08
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Advanced Biliary Cancer
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450+Anlotinib (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle ,Anlotinib capsules 12 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2450 Injection; Drug: Anlotinib hydrochloride
- Chemotherapy (Active Comparator): Capecitabine tablets combined with oxaliplatin injection or gemcitabine hydrochloride injection. Each cycle is 3 weeks.
  Interventions: Drug: Oxaliplatin injection; Drug: Capecitabine tablets; Drug: Gemcitabine hydrochloride injection

INTERVENTIONS:
Drug: TQB2450 Injection — TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle.
  Arms: TQB2450+Anlotinib
Drug: Anlotinib hydrochloride — Anlotinib capsules 12 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Arms: TQB2450+Anlotinib
Drug: Oxaliplatin injection — Oxaliplatin injection 130 mg/m2 administered IV on Day 1 of each week in 3-week cycles;
  Arms: Chemotherapy
Drug: Capecitabine tablets — Capecitabine tablets total dose 2000 mg/m2, oral twice a day from Day 1-14 of each 3- week cycles;
  Arms: Chemotherapy
Drug: Gemcitabine hydrochloride injection — Gemcitabine hydrochloride injection administered 1000 mg/m2 IV on Day 1 and Day 8 of each week in 3-week cycles.
  Arms: Chemotherapy

SUMMARY:
This study is a randomized, parallel controlled, multicentre phase III clinical trial to evaluate the efficacy and safety of TQB2450 combined with anlotinib versus chemotherapy as second-line treatment in subjects with advanced biliary cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed biliary adenocarcinoma, including intrahepatic cholangiocarcinoma (ICC), extrahepatic cholangiocarcinoma (ECC) and gallbladder cancer (GBC).

2.18 years and older,Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months;Weight ≥40 kg or BMI ≥18.5.

3. At least one measurable lesion (based on RECIST 1.1). 4. Previous first-line gemcitabine or fluorouracil-based combination chemotherapy failed.

5.Adequate laboratory indicators. 6. No pregnant or breastfeeding women, and a negative pregnancy test. 7. Understood and Signed an informed consent form.

Exclusion Criteria:

* 1. Tumor disease and medical history:

  1. Has central nervous system metastases (CNS) and/or cancerous meningitis or leptomeningeal carcinomatosis;
  2. Has other malignant tumors within 5 years;
  3. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear;
  4. Severe bone damage caused by tumor bone metastasis;
  5. Has uncontrolled and repeated drainage pleural effusion, pericardial effusion, and ascites;
  6. Partial or complete intestinal obstruction and complete biliary obstruction that cannot be relieved; 2. Previous anti-tumor therapy:

  <!-- -->

  1. Has received Anlotinib Hydrochloride Capsules, Bevacizumab Injection, and immune checkpoint inhibitors such as PD-1, PD-L1, and CTLA-4 in prior treatment;
  2. Have received anti-tumor therapy within 4 weeks before the first administration;
  3. Unalleviated toxicity ≥ grade 1 due to any previous anticancer therapy; 3.Comorbidities and medical history:

  <!-- -->

  1. Active hepatitis B or C;
  2. Kidney abnormalities;
  3. Abnormal thyroid function;
  4. Cardiovascular abnormalities;
  5. Gastrointestinal abnormalities;
  6. History of immunodeficiency;
  7. Has risk of bleeding;
  8. Uncontrollable active bacterial, fungal or viral infections;
  9. Lung diseases, such as interstitial pneumonia, obstructive lung disease, and history of symptomatic bronchospasm;
  10. Allergies to the ingredients of the study drug;
  11. Have a history of neurological or psychiatric disorders
  12. According to the researcher's point of view, other severe, acute or chronic medical or mental illnesses or laboratory abnormalities that may increase the risks associated with participating in the study, or may interfere with the interpretation of the study results;
  13. Have a history of pituitary or adrenal dysfunction
  14. Has received major surgical treatment, open biopsy, or obvious traumatic injury within 28 days before the first administration;
  15. Long-term unhealed wound or fracture;
  16. Has drug abuse history that unable to abstain from or mental disorders; 4. Has participated in other clinical trials within 30 days before the study. 5. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first administration.

      6. Pregnant or breastfeeding women. 7. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-03-18 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 40 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 24 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall response rate (ORR) | up to 24 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 24 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of response（DOR） | up to 24 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Progression-free survival at 6 months | up to 6 months
  Percentage of participants whose PFS has achieved at least 6 months.
Overall survival at 6 months | up to 6 months
  Percentage of participants whose OS has achieved at least 6 months.
Overall survival at 12 months | up to 12 months
  Percentage of participants whose OS has achieved at least 12 months.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Anhui Provincal Hospital, Hefei, Anhui
  - Beijing Chao-Yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital,Captical Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Harbin Medical University Affiliated Tumor Hospital, Harbin, Heilongjiang
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Tongji Medical College of HUST, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin